CLINICAL TRIAL: NCT01599910
Title: The Effect of Scribes in the Emergency Department
Brief Title: Scribes in the Emergency Department
Status: Withdrawn | Type: Observational
Why Stopped: Funding not received
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Steven Horng, MD, Instructor of Emergency Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: ed-scribe
Record Dates: First submitted 2012-05-15; First posted 2012-05-16 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Scribes in the Emergency Department
Keywords: Scribes; Physician Productivity; Electronic Documentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Scribes — Scribe

SUMMARY:
This study will evaluate the effect of scribes on an academic emergency department.

DETAILED DESCRIPTION:
This study will be a prospective before-after study with washout period of various performance measures before and after the implementation of ED scribes. We will also collect survey data to measure physician satisfaction and patient perception of scribes.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients during the study period
* age > 18 y/o

Exclusion Criteria:

* Patients seen during the washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult emergency department patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Time to attending chart completion | 6 months

SECONDARY OUTCOMES:
Physician productivity | 6 months
  patients / shift
Physician Reimbursement | 6 months
  RVU/hr dollars/hr
Quality of Documentation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Horng, MD, Principal Investigator — Beth Israel Deaconess Medical Center